CLINICAL TRIAL: NCT06871748
Title: Effect of a Low FODMAP Diet in Irritable Bowel Syndrome and Functional Constipation with Bloating: a Randomized Double-Blind Controlled Trial with Microbiota, Intestinal Gas, and Metabolomic Analysis
Brief Title: Effect of a Low FODMAP Diet in IBS and Functional Constipation with Bloating: a Randomized Double-Blind Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 148/2025
Record Dates: First submitted 2025-02-28; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Irritable Bowel Syndrome (IBS); Constipation - Functional; Bloating
Keywords: Irritable Bowel Syndrome (IBS); Functional Constipation; FODMAP; Microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, controlled trial investigating the effects of a low FODMAP diet compared to a high FODMAP diet in IBS and functional constipation patients with bloating. Participants will be randomly assigned to one of two dietary intervention groups for two weeks. The trial employs block randomization (block size=4). Both participants and study personnel will be blinded to the diet assignment, with identical meal appearances to maintain blinding. Outcomes include clinical symptom improvement, gut microbiota changes, gas production, and metabolomic profiles. Data will be analyzed using chi-square tests, logistic regression, and microbiome diversity metrics. This study aims to provide mechanistic insights and evidence-based dietary recommendations for managing bloating-predominant IBS and functional constipation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a double-blind design, where both participants and study personnel (including investigators, dietitians, and outcome assessors) are blinded to dietary assignments. Meals in both groups are designed to have identical appearance, texture, and calorie content, differing only in FODMAP composition to maintain blinding. Food preparation staff, who are not involved in data collection or patient interaction, will be the only personnel aware of group assignments. The randomization sequence is generated by an independent researcher who does not participate in data analysis or outcome assessment. Blinded data analysis will be conducted to prevent bias. Participants will be instructed not to discuss meal characteristics to preserve masking. This ensures objective assessment of dietary effects on bloating, microbiota composition, gas production, and metabolic profiles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low FODMAP Diet (Experimental): Participants will follow a low FODMAP diet for two weeks, consuming standardized meals with minimal fermentable carbohydrates. Meals match the high FODMAP diet in appearance to maintain blinding.
  Interventions: Other: Low FODMAP Diet
- High FODMAP Diet (Active Comparator): Participants will follow a high FODMAP diet for two weeks, consuming standardized meals with high fermentable carbohydrates. Meals match the low FODMAP diet in appearance to maintain blinding.
  Interventions: Other: High FODMAP Diet

INTERVENTIONS:
Other: Low FODMAP Diet — A standardized diet containing low levels of fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAPs), designed to reduce bloating and gastrointestinal symptoms. Meals are pre-prepared, calorie-matched, and visually identical to those in the high FODMAP group to maintain blinding. Participants will consume three main meals and one snack daily for two weeks, with adherence monitored through food diaries and photos.
  Arms: Low FODMAP Diet
Other: High FODMAP Diet — A standardized diet containing high levels of fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (FODMAPs) to assess its impact on bloating and gastrointestinal symptoms. Meals are calorie-matched and visually identical to those in the low FODMAP group to maintain blinding. Participants will consume three main meals and one snack daily for two weeks, with adherence tracked through food diaries and photos.
  Arms: High FODMAP Diet

SUMMARY:
This clinical study aims to evaluate the effects of a low FODMAP diet compared to a high FODMAP diet in patients with Irritable Bowel Syndrome (IBS) and Functional Constipation (FC) with predominant bloating. The study is a randomized, double-blind, controlled trial designed to assess whether a diet low in fermentable carbohydrates can improve bloating symptoms, gut microbiota composition, intestinal gas production, and metabolic outputs.

Patients meeting the Rome IV criteria for IBS or FC with persistent bloating will be enrolled and randomly assigned to receive either a low or high FODMAP diet for two weeks. Meals will be standardized to control FODMAPs composition, ensuring that FODMAP content is the primary variable.

The primary endpoint is the proportion of participants with a ≥30% reduction in bloating severity, measured using the Visual Analog Scale (VAS). Secondary outcomes include changes in global IBS symptoms, abdominal pain, bowel movements, stool consistency, microbiota diversity, hydrogen/methane gas production, and metabolomic profiles.

This study will contribute to the growing body of evidence supporting dietary management in disorders of gut-brain interaction (DGBI), particularly in bloating-predominant IBS and FC, and will provide insights into the mechanisms linking diet, gut microbiota, and symptom improvement.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) and Functional Constipation (FC) are chronic Disorders of Gut-Brain Interaction (DGBI) characterized by altered motility, visceral hypersensitivity, dysbiosis, and central nervous system processing abnormalities. Bloating is a challenging and distressing symptom that often persists despite standard pharmacological treatments.

The low FODMAP diet has been widely studied as a dietary approach to alleviate IBS symptoms. FODMAPs (Fermentable Oligosaccharides, Disaccharides, Monosaccharides, and Polyols) are poorly absorbed short-chain carbohydrates that increase osmolarity, promote intestinal gas production, and alter gut microbiota, leading to bloating and discomfort. Although studies support the effectiveness of the low FODMAP diet, existing research lacks controlled, blinded trials assessing its impact on bloating-specific symptoms and related physiological markers.

This study addresses these gaps by using a double-blind, controlled design with rigorously standardized meals containing well-defined FODMAP content. It will assess clinical outcomes, gut microbiota composition, gas production, and metabolomic changes to elucidate the mechanisms underlying the diet's effects.

Study Design This is a randomized, double-blind, controlled trial conducted at a single center. Participants will be assigned to receive either a low FODMAP or a high FODMAP diet for two weeks.

Participants:

Adults ≥18 years diagnosed with IBS or FC with persistent bloating based on Rome IV criteria.

Intervention:

Standardized meal plans containing either low FODMAP or high FODMAP content.

Randomization:

Computer-generated block randomization (block of 4)

Blinding:

Investigators, study staff, and participants will remain blinded to the dietary allocation.

Primary Outcome:

≥30% reduction in bloating severity on the VAS scale.

Secondary Outcomes:

Changes in global IBS symptoms (IBS-SSS) or constipation symptoms (PAC-Sym) Abdominal pain (VAS) stool frequency, and consistency (Bristol Stool Form Scale). Gut microbiota diversity and composition (16S rRNA sequencing). Intestinal gas production (hydrogen/methane breath test). Metabolomic analysis (short-chain fatty acids, urine histamine, azelaic acid). Use of rescue medications for symptom relief.

Study Procedures

Baseline Assessment:

Demographic data, medical history, and dietary habits (7-day food diary). Baseline bloating severity, stool consistency, and quality of life (IBS-QoL, PAC-QoL).

Microbiota, breath test, and metabolomic sampling.

Intervention Phase (2 Weeks):

Participants consume standardized low or high FODMAP meals (3 main meals + 1 snack/day).

Daily recording of symptoms, bowel movements, and use of rescue medications.

Follow-up Assessments:

Week 1: Phone follow-up to assess adherence and symptom progression. Week 2: Final clinical and laboratory assessments (identical to baseline). Data collection for statistical analysis comparing treatment effects.

Statistical Analysis Primary endpoint (bloating reduction) analyzed using Chi-square/Fisher's exact test.

Secondary outcomes analyzed with paired t-tests, Mann-Whitney U tests, and logistic regression.

Microbiota diversity assessed using Shannon index, beta diversity, and PERMANOVA testing.

Significance and Impact This study will provide high-quality evidence on the effectiveness of the low FODMAP diet for bloating-predominant IBS and FC, addressing critical knowledge gaps. By integrating clinical, microbiota, and metabolomic data, it will enhance understanding of diet-microbiota interactions and their role in symptom modulation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosed with Irritable Bowel Syndrome (IBS) or Functional Constipation (FC) based on Rome IV criteria
* Persistent bloating affecting daily life, with a bloating VAS score ≥4
* Stable bowel habits with Bristol Stool Form Scale (BSFS) type 3-5
* History of prior treatment with antispasmodics and/or prokinetics (allowed if dose remains stable)
* Able to comply with dietary intervention and study procedures

Exclusion Criteria:

* Prior gastrointestinal surgery (except appendectomy or cholecystectomy)
* Use of antibiotics, proton pump inhibitors (PPIs), probiotics, NSAIDs, lactulose, or metformin within the past 4 weeks
* Presence of systemic diseases affecting gut microbiota (e.g., liver cirrhosis, uncontrolled diabetes, end-stage renal disease, obesity, cancer, psychiatric disorders)
* Inability to consume study meals or follow dietary restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Bloating Severity (VAS) | Baseline to 2 weeks (End of Intervention)
  The primary outcome is the change in bloating severity, measured using the Visual Analog Scale (VAS). The VAS score ranges from 0 (no bloating) to 10 (severe bloating), with higher scores indicating worse bloating symptoms. Participants will record daily bloating scores throughout the intervention period. The proportion of participants achieving a ≥30% decrease in bloating severity from baseline will be analyzed.

SECONDARY OUTCOMES:
Reduction in Global IBS Symptoms (IBS-SSS) | Baseline to 2 weeks
  Change in IBS Symptom Severity Score (IBS-SSS) from baseline, assessing overall IBS symptom burden, abdominal pain, bloating, and bowel habit changes. The IBS-SSS scale ranges from 0 to 500, with higher scores indicating more severe IBS symptoms.
Change in Abdominal Pain (VAS) | Baseline to 2 weeks
  Change in abdominal pain severity, measured using the Visual Analog Scale (VAS). The VAS scale ranges from 0 (no pain) to 10 (severe pain), with higher scores indicating worse pain severity. Participants will record daily pain scores, and the difference between baseline and post-intervention scores will be analyzed.
Change in Stool Frequency and Consistency | Baseline to 2 weeks
  Change in bowel movement frequency and stool consistency, assessed using the Bristol Stool Form Scale (BSFS).
  Stool frequency will be recorded as the number of bowel movements per day.
  Stool consistency will be graded using the BSFS scale (1-7):
  1-2: Hard stools (constipation) 3-4: Normal stools 5-7: Loose stools (diarrhea) Higher BSFS scores indicate looser stool consistency. The difference between baseline and post-intervention values will be analyzed.
Changes in Gut Microbiota Composition | Baseline to 2 weeks
  Alterations in gut microbiota diversity and abundance (16S rRNA sequencing).
Change in Hydrogen Gas Production (Lactulose Breath Test) | Baseline to 2 weeks
  Change in exhaled hydrogen (H₂) levels, measured via lactulose breath test in parts per million (ppm). Higher hydrogen levels indicate increased fermentation by colonic microbiota.
Change in Methane Gas Production (Lactulose Breath Test) | Baseline to 2 weeks
  Change in exhaled methane (CH₄) levels, measured via lactulose breath test in parts per million (ppm). Elevated methane levels are associated with slow colonic transit and constipation.
Use of Rescue Medications | Baseline to 2 weeks
  Frequency and dosage of antispasmodics, prokinetics, or laxatives used for symptom relief.
Change in Psychological Symptoms (DASS-21) | Baseline to 2 weeks
  Change in Depression, Anxiety, and Stress Scores (DASS-21), a validated self-reported scale measuring psychological distress. The DASS-21 consists of three subscales:
  Depression (0-21) Anxiety (0-21) Stress (0-21) Each subscale score ranges from 0 (normal) to 21 (severe symptoms), with higher scores indicating greater psychological distress. The total score is calculated by summing individual subscale scores.
Change in Quality of Life (IBS-QoL / PAC-QoL) | Baseline to 2 weeks
  Change in IBS-specific Quality of Life (IBS-QoL) score, which assesses the impact of IBS on daily activities, emotional well-being, and social functioning.
  The IBS-QoL score ranges from 0 to 100, with higher scores indicating better quality of life.
Patient Satisfaction with Treatment | Baseline to 2 weeks
  Overall treatment satisfaction, measured using a Visual Analog Scale (VAS) ranging from 0 to 10:
  0 = Completely Dissatisfied 10 = Completely Satisfied Higher scores indicate greater satisfaction with treatment. The difference between baseline and post-intervention scores will be analyzed.
Change in Patient-Reported Constipation Symptoms (PAC-SYM) | Baseline to 2 weeks
  Change in Patient Assessment of Constipation-Symptoms (PAC-SYM) score, evaluating constipation-related symptoms, including stool consistency, discomfort, and straining. The PAC-SYM scale ranges from 0 to 48, with higher scores indicating worse constipation symptoms.
Change in Short-Chain Fatty Acids (SCFAs) Levels | Baseline to 2 weeks
  Change in fecal short-chain fatty acids (SCFAs), including acetic acid, propionic acid, and butyric acid, measured in μmol/g stool. Higher SCFA levels indicate greater microbial fermentation activity.
Change in Urine Histamine Levels | Baseline to 2 weeks
  Change in urine histamine concentration, measured in μg/mL urine, assessing histamine metabolism related to gut inflammation and microbiota activity. Higher levels indicate increased histamine production.
Change in Urine Azelaic Acid Levels | Baseline to 2 weeks
  Change in urine azelaic acid concentration, measured in μg/mL urine, assessing microbial metabolic changes associated with gut dysbiosis and inflammation. Higher levels indicate altered microbial metabolism.
Change in Constipation-Specific Quality of Life (PAC-QoL) | Baseline to 2 weeks
  Change in Patient Assessment of Constipation-Quality of Life (PAC-QoL) score, evaluating the impact of constipation on daily life, physical discomfort, psychological well-being, and social aspects.
  The PAC-QoL score ranges from 0 to 100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Monthira Maneerattanaporn, MD, Study Director — Mahidol University Faculty of Medicine Siriraj Hospital; Tanawat Geeratragool, MD, Principal Investigator — Mahidol University Faculty of Medicine Siriraj Hospital; Somchai Leelakusolvong, MD, Study Chair — Mahidol University Faculty of Medicine Siriraj Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drossman DA, Tack J. Rome Foundation Clinical Diagnostic Criteria for Disorders of Gut-Brain Interaction. Gastroenterology. 2022 Mar;162(3):675-679. doi: 10.1053/j.gastro.2021.11.019. Epub 2021 Nov 19. No abstract available. PMID 34808139
- [Background] Camilleri M. Diagnosis and Treatment of Irritable Bowel Syndrome: A Review. JAMA. 2021 Mar 2;325(9):865-877. doi: 10.1001/jama.2020.22532. PMID 33651094
- [Background] Andrews CN, Sidani S, Marshall JK. Clinical Management of the Microbiome in Irritable Bowel Syndrome. J Can Assoc Gastroenterol. 2020 Jan 4;4(1):36-43. doi: 10.1093/jcag/gwz037. eCollection 2021 Feb. PMID 33644675
- [Background] Varney J, Barrett J, Scarlata K, Catsos P, Gibson PR, Muir JG. FODMAPs: food composition, defining cutoff values and international application. J Gastroenterol Hepatol. 2017 Mar;32 Suppl 1:53-61. doi: 10.1111/jgh.13698. PMID 28244665
- [Background] Muir JG, Shepherd SJ, Rosella O, Rose R, Barrett JS, Gibson PR. Fructan and free fructose content of common Australian vegetables and fruit. J Agric Food Chem. 2007 Aug 8;55(16):6619-27. doi: 10.1021/jf070623x. Epub 2007 Jul 11. PMID 17625872